CLINICAL TRIAL: NCT03757078
Title: Prospective Multicenter Non-interventional Study of Fluocortolone + Lidocaine Formulation in Patients With Acute Hemorrhoids to Evaluate Changes in Symptoms Severity During the Course of Treatment
Brief Title: Study to Find Out How Symptoms Severity Changes During the Standard Course of Treatment With the Cream Relief Pro and Suppositories Relief Pro (Active Ingredients Are Fluocortolone + Lidocaine) in Patients Suffering From Twisted and Bulging Veins in the Rectal Area (Acute Hemorrhoids)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20364
Record Dates: First submitted 2018-10-26; First posted 2018-11-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Acute Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute hemorrhoids: Patients with acute hemorrhoids of 1-2 stage were prescribed Fluocortolone + Lidocaine by a physician. No drug will be provided to Patient by the Investigator, only prescription order, based on International Nonproprietary name (Fluocortolone + Lidocaine)
  Interventions: Drug: Relief Pro cream; Drug: Relief Pro rectal suppositories

INTERVENTIONS:
Drug: Relief Pro cream — Relief Pro cream:1.0 mg/gm Fluocortolone + 20 mg/gm Lidocaine; Administration according to clinical practice.
Drug: Relief Pro rectal suppositories — Relief Pro rectal suppositories: 1.0 mg Fluocortolone + 40 mg Lidocaine; Administration according to clinical practice

SUMMARY:
In this study researcher wanted to learn more about the changes of biggest twisted and bulging veins in the rectal area (hemorrhoids) and changes of symptoms during a treatment period with the cream Relief Pro and suppositories Relief Pro. The study collected information on the treatment satisfaction of patients and their physicians with the prescribed treatment by using questionnaires. There were 3 visits at the physician's clinic for this study: one initial visit and 2 follow-up visits over a period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male & female patients 18 to 65 years old;
* Patients with acute hemorrhoids 1 and 2 stage (with thrombosis (external, internal, mixed), including cases with bleeding);
* Prescription of fluocortolone + lidocaine as a part of routine clinical practice.

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice;
* Hemorrhoid with stage ˃ II;
* Contraindications for use of Relief PRO in the approved product label;
* Anemia and/or severe/profuse hemorrhoid bleeding;
* Surgery in perianal region in anamnesis;
* Concomitant treatment with antibiotics/antiseptics, antithrombotics, antineoplastic and/or immunosuppressant;
* Inflammatory bowel disease;
* Hepatic diseases in severe and acute stages;
* Colorectal cancer;
* Purulent-inflammatory diseases of the perianal region and anal canal;
* Chronic pulmonary diseases in severe and acute stages.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with acute hemorrhoids from Russia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Severity of pain (VAS: Visual Analogue Scale) | Up to 14 days
  Pain was measured on a Visual Analogue Scale (VAS) from 0 (No Pain) to 10 (Maximal Pain).
Severity of bleeding (according to 4-point Likert scale) | Up to 14 days
  4-point Likert scale consisting of: 1 (None), 2 (Minimal), 3 (Moderate) and 4 (Significant).
Severity of pruritus (according to 4-point Likert scale) | Up to 14 days
Severity of swelling (according to 4-point Likert scale) | Up to 14 days
Severity (amount) of discharge (according to 4-point Likert scale) | Up to 14 days
Severity of sense of discomfort (according to 4-point Likert scale) | Up to 14 days
Overall patient satisfaction with treatment (according to 5-point Likert scale) | Up to 14 days
  Likert scale: 1 (Very satisfied), 2 (Satisfied), 3 (Neither satisfied nor dissatisfied), 4 (Dissatisfied) and 5 (Very dissatisfied).
Time to onset of analgesic effect after the first use of the drug | Up to 14 days
Duration of analgesic effect after the first use of the drug | Up to 14 days
Patient's adherence to recommendations of the Investigator by PRO | Up to 14 days
  PRO: Patient Reported Outcome
Information obtained in the course of questioning about the consumer properties of the study product by PRO | Up to 14 days
Severity of hemorrhoids symptoms according to the Sodergren score | Up to 14 days
  Standardized answer options are given (4 and 5 Likert boxes) and each question gets a score from 0 to 4.
Size of the largest hemorrhoid node measured during a routine examination | Up to 14 days
Severity of swelling when assessed as part of routine examination (according to 4-point Likert scale) | Up to 14 days
Severity of bleeding when assessed as part of routine examination (according to 4-point Likert scale) | Up to 14 days
Amount of ReliefPro used based on information provided by the patient to the Investigator | Up to 14 days
Overall satisfaction of Investigator with treatment with Relief Pro according Likert scale from 1 to 5 points as measured on Visits 2 and 3 | Up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Center of Coloproctology, Moscow, Russia

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/